CLINICAL TRIAL: NCT00002267
Title: Rifabutin Therapy for the Prevention of Mycobacterium Avium Complex (MAC) Bacteremia in AIDS Patients With CD4 Counts = or < 200: A Double-Blind, Placebo-Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pharmacia (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 048B; 087027-999
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1992-03

CONDITIONS: Mycobacterium Avium-intracellulare Infection; HIV Infections
Keywords: Rifabutin; AIDS-Related Opportunistic Infections; Mycobacterium avium-intracellulare Infection; Acquired Immunodeficiency Syndrome; Antitubercular Agents
MeSH Terms: conditions — Mycobacterium avium-intracellulare Infection; HIV Infections; AIDS-Related Opportunistic Infections; Acquired Immunodeficiency Syndrome | interventions — Rifabutin

INTERVENTIONS:
Drug: Rifabutin

SUMMARY:
The primary objective of this trial is to assess the safety and the relative benefit of rifabutin monotherapy in preventing or delaying the incidence of Mycobacterium avium complex (MAC) bacteremia in AIDS patients with CD4 counts less than or equal to 200, as compared to placebo, and to assess if survival is prolonged in patients who receive rifabutin prophylaxis.

ELIGIBILITY:
Inclusion Criteria

Patients must have the following:

* Diagnosis of AIDS with a case defining infection other than Mycobacterium avium complex (MAC).
* Written informed consent obtained, which must include a statement that treatment may involve risks to the embryo or fetus, which are currently unforeseeable, if the subject becomes pregnant.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Known hypersensitivity to rifabutin, rifampin, other rifamycins, zidovudine or didanosine (ddI).
* Previous or current infection due to Mycobacterium avium complex (MAC) disease as evaluated by two successive blood cultures and two successive stool cultures taken within 14 days prior to study initiation.

Concurrent Medication:

Excluded:

* Antiretroviral agents other than zidovudine (AZT).
* Didanosine (ddI).
* Antimycobacterial therapy.
* Rifampin.
* Isoniazid.
* Clofazimine.
* Ethambutol.
* Cycloserine.
* Ethionamide.
* Amikacin.
* Ciprofloxacin.
* Streptomycin.
* Other investigational drugs.
* If antimicrobial therapy is required to treat bacterial infections (= or < 14 days), Adria Laboratories must be contacted prior to initiation of therapy.

Patients with the following are excluded:

* Known hypersensitivity to rifabutin, rifampin, other rifamycins, zidovudine (AZT), or didanosine (ddI).
* Previous or current Mycobacterium avium complex (MAC) infection.
* Perceived patient unreliability or unavailability for frequent monitoring.

Prior Medication:

Excluded within 4 weeks of study entry:

* Antiretroviral agents other than zidovudine (AZT) or didanosine (ddI).
* Antimycobacterial therapy.
* Rifampin.
* Isoniazid.
* Clofazimine.
* Ethambutol.
* Cycloserine.
* Ethionamide.
* Amikacin.
* Ciprofloxacin.

Required:

* Zidovudine (AZT).
* Antipneumocystis prophylactic therapy.

Required for at least 4 weeks prior to study entry:

* Zidovudine (AZT) or didanosine (ddI).
* Antipneumocystis prophylaxis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750

CONTACTS AND LOCATIONS:
Locations (43):
- United States (31):
  - Maricopa County Med Ctr, Phoenix, Arizona
  - East Bay AIDS Ctr, Berkeley, California
  - Pacific Oaks Med Group, Beverly Hills, California
  - AIDS Community Research Consortium, Redwood City, California
  - HIV Research Group, San Diego, California
  - Dr Larry A Waites, San Francisco, California
  - Saint Francis Mem Hosp / HIV Care, San Francisco, California
  - Dr Marcus Conant, San Francisco, California
  - San Francisco Veterans Administration Med Ctr, San Francisco, California
  - Dr Marshall Kubota, Santa Rosa, California
  - Dr Jeffrey Galpin, Tarzana, California
  - Miami Veterans Administration Med Ctr, Miami, Florida
  - Community Research Initiative of South Florida, Miami, Florida
  - Northwestern Univ Med School, Chicago, Illinois
  - AIDS Research Alliance - Chicago, Chicago, Illinois
  - Tulane Univ School of Medicine, New Orleans, Louisiana
  - Comprehensive AIDS Alliance of Detroit / Harper Hosp, Detroit, Michigan
  - Univ of Minnesota, Minneapolis, Minnesota
  - St Paul Ramsey Med Ctr, Saint Paul, Minnesota
  - Univ of Nevada / Veterans Administration Med Ctr, Reno, Nevada
  - North Jersey Community Research Initiative, Newark, New Jersey
  - Univ of New Mexico Hlth Sciences Ctr / Dept of Med, Albuquerque, New Mexico
  - Dr Donald Romig, Sante Fe, New Mexico
  - Albany Veterans Administration, Albany, New York
  - AIDS Services Erie County Med Ctr, Buffalo, New York
  - Community Health Network, Rochester, New York
  - Buckley Braffman Stern Med Associates, Philadelphia, Pennsylvania
  - Thomas Jefferson Med College, Philadelphia, Pennsylvania
  - Dr Alfred F Burnside Jr, Columbia, South Carolina
  - Infectious Disease Physicians Inc, Annandale, Virginia
  - Milwaukee County Med Complex, Milwaukee, Wisconsin
- Canada (12):
  - Univ of Calgary Health Science Ctr, Calgary, Alberta
  - Univ of Alberta/Division of Inf Dis/Dept of Med, Edmonton, Alberta
  - Saint Paul's Hosp, Vancouver, British Columbia
  - Victoria Gen Hosp, Halifax, Nova Scotia
  - McMaster Univ Med Ctr, Hamilton, Ontario
  - Ottawa Gen Hosp, Ottawa, Ontario
  - Mount Sinai Hosp, Toronto, Ontario
  - Saint Michael's Hosp, Toronto, Ontario
  - Sunnybrook Health Science Ctr, Toronto, Ontario
  - Dr Emil Toma / Hotel Dieu de Montreal, Montreal, Quebec
  - Montreal Chest Institute, Montreal, Quebec
  - Montreal Gen Hosp, Montreal, Quebec

REFERENCES:
- [Background] Dautzenberg B, Castellani P, Pellegrin JL, Vittecoq D, Truffot-Pernot C, Pirotta N, Sassella D. Early bactericidal activity of rifabutin versus that of placebo in treatment of disseminated Mycobacterium avium complex bacteremia in AIDS patients. Antimicrob Agents Chemother. 1996 Jul;40(7):1722-5. doi: 10.1128/AAC.40.7.1722. PMID 8807071
- [Background] Moore RD, Chaisson RE. Survival analysis of two controlled trials of rifabutin prophylaxis against Mycobacterium avium complex in AIDS. AIDS. 1995 Dec;9(12):1337-42. doi: 10.1097/00002030-199512000-00006. PMID 8605053